CLINICAL TRIAL: NCT05151406
Title: Myths and Misconceptions About HSCT in a Limited Resource Region: Current Situation and Future Directions
Brief Title: Myths and Misconceptions About HSCT in a Limited Resource Region
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esmat Sayed Abd elmageed, assistant professor of medical surgical nursing, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Esmat19
Record Dates: First submitted 2021-10-12; First posted 2021-12-09 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Intervention Model Description: An intervention Quasi Experimental study design (pre/post-test)
Who Masked: Participant
Masking Description: coding of data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- medical students (Active Comparator): 5th year undergraduate medical students
  Interventions: Other: educational program
- nursing students (Active Comparator): 4th year undergraduate nursing students
  Interventions: Other: educational program

INTERVENTIONS:
Other: educational program — The needed knowledge about hematopoietic stem cell transplantation in a trial to correct their myths and misconceptions about this type of treatment. The educational pamphlet included three theoretical parts: bone marrow transplantation, bone marrow donation, and stem cells banking

SUMMARY:
This study aimed to assess myths and misconceptions about hematopoietic stem cell transplantation, among students of medical colleges and to evaluate the value of an educational program in correcting those misconceptions. 218 undergraduate medical and nursing students included in this study. An intervention Quasi Experimental study design (pre/post-test) was used for this work.

DETAILED DESCRIPTION:
This study aimed to assess myths and misconceptions about hematopoietic stem cell transplantation, among students of medical colleges and to evaluate the value of an educational program in correcting those misconceptions. The last aim was to detect further needs for advancement of health education about bone marrow transplantation at Assiut University.

Study subjects: two groups, Group 1: 5th year undergraduate medical students(118 students), Group 2: 4th year undergraduate nursing students(100 students). Each group were randomly selected . Both groups 1 and 2 assumed to have knowledge about BMT from their study courses, also they represent a sector from the general population that could be involved in a BMT team in their future career. this work that was conducted at Assiut University Faculties of Medicine and Nursing at Assiut Governorate during the period from July 2019 to May 2020. The subject's inclusion criteria were:

* Willingness to participate in the study
* Good ECOG performance status
* Intact physical and mental health

And the Exclusion criteria were:

* HSCT team
* Drug users

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate in the study
* Good ECOG performance status
* Intact physical and mental health

Exclusion Criteria:

* HSCT team
* Drug users

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 218 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Assess myths and misconceptions about hematopoietic stem cell transplantation using structured questionnaire about misconceptions and willingness regarding hematopoietic stem cell transplantation | one session for medical students and one session for nursing students, each session will take up to 1 hour
  5th year undergraduate medical students and 4th year undergraduate nursing students will be asked about their misconceptions about hematopoietic stem cell transplantation including bone marrow transplantation, bone marrow donation, and stem cell banking.

SECONDARY OUTCOMES:
evaluate the value of an educational program by using structured questionnaire (Part II and Part III) willingness regarding hematopoietic stem cell transplantation and misconceptions about hematopoietic stem cell transplantation | one session for medical students and one session for nursing students, each session will take up to 1 hour
  the educational program corrects myths and misconceptions about hematopoietic stem cell transplantation of the study sample and increases their willingness regarding hematopoietic stem cell transplantation

OTHER OUTCOMES:
detect further needs for advancement of health education by using structured questionnaire (Part II and Part III) willingness regarding hematopoietic stem cell transplantation and misconceptions about hematopoietic stem cell transplantation | one session for medical students and one session for nursing students, each session will take up to 1 hour
  the educational program corrects myths and misconceptions about hematopoietic stem cell transplantation of the study sample and increases their willingness regarding hematopoietic stem cell transplantation which enhance the needs for advancement of health education about bone marrow transplantation at Assiut University.

CONTACTS AND LOCATIONS:
Overall Officials: safaa a Abd-elsatar, Assist prof, Principal Investigator — faculty of medicine
Locations (1):
- Faculty of medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
protocol
Supporting Information: Study Protocol
Time Frame: 12/8/2021
Access Criteria: protocol

REFERENCES:
- [Derived] Khaled SAA, Elzembely MM, Soliman AMA, Shwakat N, Rafaat N, Malek MA, Abdelmageed ES. Effective and Elaborative Induction Program for Mitigating Myths and Misconceptions Linked to Hematopoietic Stem Cell Transplantation in a Resource Limited Setting. Indian J Hematol Blood Transfus. 2023 Oct;39(4):598-609. doi: 10.1007/s12288-023-01634-5. Epub 2023 Mar 16. PMID 37786824